CLINICAL TRIAL: NCT04489719
Title: The Impact of DNA Repair Pathway Alterations Identified by Circulating Tumor DNA on Sensitivity to Radium-223 in Bone Metastatic Castration-Resistant Prostate Cancer
Brief Title: Impact of DNA Repair Pathway Alterations on Sensitivity to Radium-223 in Bone Metastatic Castration-resistant Prostate Cancer
Status: Recruiting | Type: Observational
Sponsor: University of Washington (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: RG1006011; NCI-2020-04699 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10370 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2020-07-23; First posted 2020-07-28 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Castration-Resistant Prostate Carcinoma; Metastatic Malignant Neoplasm in the Bone; Metastatic Prostate Carcinoma; Stage IVB Prostate Cancer AJCC v8
Keywords: Prostate
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Specimen Handling; radium Ra 223 dichloride

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observational (biospecimen collection): Patients receive standard of care radium Ra 223 dichloride given by IV bolus every 4 weeks for up to 6 cycles. Patients undergo collection of blood every 1-3 months during radium Ra 223 dichloride treatment.
  Interventions: Procedure: Biospecimen Collection; Other: Questionnaire Administration; Drug: Radium Ra 223 Dichloride

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Other: Questionnaire Administration — Ancillary studies
Drug: Radium Ra 223 Dichloride — Given IV
  Other Names: Alpharadin; BAY 88-8223; BAY88-8223; Radium 223 Dichloride; RADIUM RA-223 DICHLORIDE; Radium-223 Dichloride; Xofigo

SUMMARY:
This study investigates how well radium-223 works in treating patients with castration-resistant prostate cancer than has spread to the bones (bone metastases). Prostate cancer is the most common cancer in men and the second leading cause of cancer death. Furthermore, many men with notably advanced disease have been found to have abnormalities in DNA repair. The purpose of this research is to study the role of a DNA repair pathway in prostate cancer, specifically in response to administration of radium-223, an FDA-approved drug known to cause DNA damage to cancerous cells. Understanding how defects in the DNA repair pathway affects radium-223 treatment of prostate, may help doctors help plan effective treatment in future patients.

DETAILED DESCRIPTION:
OUTLINE:

Patients receive standard of care radium Ra 223 dichloride given by intravenous (IV) bolus every 4 weeks for up to 6 cycles. Patients undergo collection of blood every 1-3 months during radium Ra 223 dichloride treatment.

After completion of study, patients are followed up every 3 months for up to 5 years from the date of treatment completion.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be >= 18 years of age
* Patient must have histopathologic diagnosis of prostate cancer
* Patient must have castration-resistant prostate cancer
* Patient must have radiographic evidence of bone metastasis
* Patients must be symptomatic from prostate cancer
* Patient must have plans to undergo treatment with radium-223
* Patient must have a PSA level >= 10 ng/mL
* Patient must have castrate testosterone levels demonstrated within the last 3 months prior to screening
* Patient must have anticipated survival > 3 months
* Patient must be willing and able to authorize consent
* Patient must be willing and able to comply with the protocol, including follow-up visits

Exclusion Criteria:

* Patient must not have visceral metastasis
* Patients on regimens of radium-223 in combination with other antineoplastic agents are excluded

  * Bone-targeted only therapy (e.g. denosumab or zoledronic acid) will be allowed
* Patients who have received prior radium-223
* Patients who have received prior platinum containing chemotherapy
* Absolute neutrophil count (ANC) < 1.5 x 10^9/L
* Hemoglobin (HB) < 9 g/dL
* Platelets (PLT) < 100 x 10^9/L
* Any condition which, in the investigator's opinion, makes the subject unsuitable for trial participation

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with mCRPC with bone metastases who are undergoing treatment with radium-223
Sampling Method: Non-Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2021-04-16 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2029-08-01 (Estimated)

PRIMARY OUTCOMES:
Response rate | Up to 1 year
  Response will be defined as having one or both of the following: confirmed prostate specific antigen (PSA) decline of >= 30% from baseline AND/OR confirmed alkaline phosphatase (ALP) decline >= 30% from baseline. Response is evaluated throughout the course of treatment until the post-radium-223 end of treatment laboratory studies. Confirmation of response by PSA and/or ALP requires a second consecutive value obtained >= 2 weeks after the first with sustained >= 30% decline. Characterization of response rate to radium-223 in the DRD patient population will be assessed by binomial proportion with Clopper-Pearson exact 2-sided 95% confidence intervals.

SECONDARY OUTCOMES:
Response rate | Up to 1 year
  Comparison of treatment response (outcome/dependent variable) between cases and controls will be assessed using multivariate logistic regression modelling adjusting for secondary variables as appropriate. Risk estimates will include odds ratios with 95% confidence intervals.
Response rate in those with previous PARP inhibitor therapy | Up to 1 year
  A multivariate logistic model with PARP inhibitor status as a secondary independent variable and a sensitivity analysis excluding those exposed to PARP inhibitors.
Overall survival | Up to 5 years
  Survival by DRD status will be illustrated using univariate Kaplan-Meier curves. Additionally, Cox-PH model adjusting for age, Eastern Cooperative Oncology Group (ECOG) performance status, Gleason grade score, baseline ALP, PSA, hemoglobin (HB), and lactate dehydrogenase (LDH) will be performed. This analysis may be limited by expected small number of events, thus it may be limited to raw reporting of events by DRD status.
Number of radium Ra 223 dichloride | Up to 6 months
Pain assessment | Up to 1 year
  Assessed via Brief Pain Inventory survey
Analgesic usage | Up to 1 year
Quality of life (FACT-P survey) | Up to 1 year
  Assessed via FACT-P quality of life survey
Incidence of adverse events | Up to 1 year
  To access risk of adverse events by DRD status, 2 logistic models will be used. The first will classify the dependent variable as an adverse event while the second model will classify the dependent variable as an adverse event < grade 3.
Response rate | Up to 1 year
  Investigate whether response rates by DRD versus non-DRD patients are modified by germline or somatic alteration status of DNA repair pathways.

CONTACTS AND LOCATIONS:
Overall Officials: Evan Y. Yu, MD, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (4):
- United States (4):
  - Johns Hopkins University, Baltimore, Maryland
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington
  - University of Wisconsin-Madison, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No